CLINICAL TRIAL: NCT00749736
Title: The Role of Vitamin D in Immune Function in Patients With CKD Stages 3 and 4.
Brief Title: The Role of Vitamin D in Immune Function in Patients With Chronic Kidney Disease (CKD) Stages 3 and 4.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0707-04
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease
Keywords: vitamin D; determine; normal; intrapatient; interpatient; variability; measures; immune system
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cholecalciferol; 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 4000 IU of cholecalciferol per day
  Interventions: Dietary Supplement: cholecalciferol
- 2 (Active Comparator): 1 mcg of doxercalciferol per day.
  Interventions: Dietary Supplement: doxercalciferol
- 3 (Placebo Comparator): placebo for six months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 4000 IU of cholecalciferol per day
  15 patients will be enrolled in each arm.
  Arms: 1
Dietary Supplement: doxercalciferol — 1 mcg of doxercalciferol per day
  Arms: 2
Dietary Supplement: placebo — placebo for 6 months; with stratification based on stage of CKD by modified MDRD formula.
  15 patients will be enrolled in each arm.
  Arms: 3

SUMMARY:
Patients with chronic kidney disease (CKD) are commonly deficient in vitamin D, with low levels of both calcidiol (25 hydroxy vitamin D) and calcitriol (1,25-hydroxy vitamin D). Patients with CKD are also known to have abnormalities in their immune cells, increased susceptibility to infection and increased prevalence of malignancies. In patients without kidney disease, repletion of vitamin D appears to help some immune mediated diseases. Thus it is logical that patients with CKD who are vitamin D deficient may benefit from repletion of vitamin D, in either its native form (cholecalciferol/ergocalciferol) or in the form of calcitriol or its analogues. However, no interventional data demonstrates that repletion positively impacts immune status in CKD patients. To test this hypothesis, a large interventional study will be required. However, prior to conducting this study, several important steps are needed. The present proposal aims to generate the necessary data to appropriately plan and conduct a future multi center interventional study. Specifically, we will examine the following specific aims in a population of CKD stage 3 and 4 subjects from Indiana University Affiliated Nephrology Clinics and determine

1. if abnormalities in immune cells and immune blood tests are related to abnormalities in vitamin D.
2. how reproducible these changes are on repeat testing and
3. if repletion of vitamin D changes these cells and immune blood tests in a small pilot study.

ELIGIBILITY:
Inclusion Criteria:

* no administration of any form of vitamin D supplement or therapy in the last 60 days except for that in a multi vitamin
* Hgb >10 mg/dl
* able to sign informed consent
* CKD stage 3 (GFR 30-59ml/min) or stage 4 (GFR 15-29ml/min)
* iPTH <70pg/ml for stage 3 or iPTH <110pg/ml for stage 4
* calcidiol levels < or +20ng/ml

Exclusion Criteria:

* initial corrected Calcium >9.7mg/dl
* initial serum Phosphorus >5.0mg/dl
* initial standardized blood pressure of >160/100
* history of significant liver disease or cirrhosis
* anticipated requirement for dialysis in 6 months
* malabsorption, severe chronic diarrhea, or ileostomy
* no calcimimetic or active vitamin D therapy 60 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the change in CD4+/CD8+ ratio and other flow cytometry parameters based on the results of Aims 1 and 2, TH1/TH2 cytokine profile, and conversion from anergic to reactive skin testing. | 6 months from baseline visit

SECONDARY OUTCOMES:
A change in mean blood pressure from one week of ambulatory measures, random protein/creatinine ratio, and differences in muscle strength by timed up and go test, and measures of quality of life using the SF36 forms. | 6 months from baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Moe, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States